CLINICAL TRIAL: NCT05771688
Title: Fetoscopic Endoluminal Tracheal Occlusion for Severe Left-sided Congenital Diaphragmatic Hernia
Brief Title: Fetoscopic Endoluminal Tracheal Occlusion
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1397678; 2021-055
Record Dates: First submitted 2023-02-16; First posted 2023-03-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Hernia, DIaphragmatic, Congenital
MeSH Terms: conditions — Hernia, Diaphragmatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- FETO therapy (Experimental): FETO therapy
  Interventions: Device: FETO therapy

INTERVENTIONS:
Device: FETO therapy — placement of FETO prior to 29 weeks 6 days GA; and removal of the FETO device no later than 35 weeks and 6 days
  Other Names: Fetoscopic Endoluminal Tracheal Occlusion; GOLDBALLOON; BALTACCI

SUMMARY:
This is a single site pilot trial to study the feasibility of Fetoscopic Endoluminal Tracheal Occlusion (FETO) therapy in the most severe group of fetuses with congenital diaphragmatic hernia (CDH) at Midwest Fetal Care Center, a collaboration between Allina Health and Children's Minnesota. This procedure aims to increase fetal lung volume before birth and improve survival after birth. This study will enroll 10 pregnant people and their baby who meet study criteria.

DETAILED DESCRIPTION:
This is a single site pilot trial to assess the feasibility and safety of treating the most severe group of fetuses with left CDH with Fetal Endoluminal Tracheal Occlusion (FETO) using the Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100) at Midwest Fetal Care Center (MWFCC), a collaboration between Allina Health and Children's MN.

Congenital Diaphragmatic Hernia (CDH) is a condition in which a hole in the baby's diaphragm allows the abdominal organs to move into the chest and limit lung growth. The goal of the FETO device is to block the airway with a balloon-type device, allowing fluid to build up in the lungs and help the unborn baby's lungs grow. Bigger lungs may improve the baby's quality of life. The rationale for fetal therapy in severe CDH is to improve fetal lung growth and therefore neonatal survival.

The study will enroll pregnant women that meet study criteria, and their baby. The mother-fetus participant will undergo one procedure for placement of FETO before gestational age 29 weeks 6 days; and a second procedure for removal of the FETO device. The timing for removal of FETO is no later than 35 weeks and 6 days. After delivery, routine care of the baby with CDH will occur within the Children's MN NICU.

ELIGIBILITY:
Inclusion Criteria:

1. A subject is defined as a female (18 years or older) who is pregnant.
2. The pregnancy must be a singleton pregnancy.
3. The CDH must be left-sided.
4. The CDH must be severe (Observed to Expected Lung to Head Ratio - O/E LHR - < 25% from U/S measurements).
5. No associated lethal anomalies (other than the CDH), no pathogenic variants on microarray, and no pathologic findings on karyotype.
6. Fetal echocardiogram with changes expected with CDH and no major structural cardiac defects.
7. Gestational age at time of balloon placement between and including 27 weeks 0 days and 29 weeks 6 days.
8. Cervix length longer than 20 mm at pre-balloon placement evaluation.
9. Acceptance of responsibility to stay locally (within 15 minutes) of MWFCC and Children's Minnesota - Minneapolis.
10. Written consent must be obtained.
11. Must meet psychosocial criteria including appropriate family/friend support during stay with balloon in place (cannot stay without additional helper), no current illicit drug use, no over-the-counter drug abuse, and no ineffectively treated DSM-IV diagnoses.

Exclusion Criteria:

1. Twin or higher order gestation
2. Not able to consent
3. Right-sided or bilateral CDH
4. Additional fetal or genetic abnormalities that would impact care after delivery or be known to have an impact on outcome
5. Maternal isoimmunization or neonatal alloimmune thrombocytopenia
6. Balloon not able to be placed prior to 30 weeks gestation
7. CDH O/E LHR 25% or greater
8. Maternal factors precluding safe fetal surgery (maternal cardiac findings not safe for anesthesia, maternal morbid obesity precluding safe usage of the equipment required for entry into the uterus, spontaneous preterm delivery prior to 36 weeks)
9. Maternal HIV, Hepatitis B with positive surface antigen, Hepatitis C with presence of virus in maternal blood due to risks of fetal transmission during procedures
10. Short cervix (20 mm or less)
11. History of incompetent cervix or uterine anomaly predisposing to preterm labor
12. Significant placental abnormalities (abruption, chorioangioma, accrete) known at the time of enrollment and/or surgery
13. History of natural rubber latex allergy
14. No safe or feasible fetoscopic approach to balloon placement
15. Inability to relocate to within 15 minutes of MWFCC/Children's Minnesota

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Successful placement of Balt Goldbal2 balloon | Prior to 29 weeks 6 days Gestational Age (GA)
  Successful completion of balloon insertion in fetuses with severe CDH defined as direct visualization of balloon above the carina at the time of FETO procedure.
Successful removal of Balt Goldbal2 balloon | Prior to 35 weeks 6 days GA
  Removal of the balloon

SECONDARY OUTCOMES:
Change in fetal lung growth | Immediately after intervention (device removal)
  Prenatal ultrasound will measure the observed-to-expected lung to head ratio (o/e LHR) at weekly visits while the balloon is in place and after balloon removal. Fetal lung growth will be calculated as the difference between the o/e LHR pre-balloon placement and the o/e LHR after balloon removal.
Gestational age at delivery | Measured at time of delivery
  Gestational age at delivery will be recorded.
Infant survival | Birth - 24 months
  Infant survival will be recorded from delivery to NICU discharge, and at 6, 12, and 24 months of age
Number of infants requiring extra corporeal membrane oxygenation (ECMO) support | Birth to 6 months
  Use of ECMO will be collected from medical chart review.
Number of infants requiring tracheostomy while in the NICU | up to 2 years of age
  Tracheostomy information will be collected from medical chart review.
Number of infants requiring home oxygen support upon discharge from the NICU | up to 2 years of age
  Oxygen support will be collected from medical chart review.
Time to pulmonary hypertension resolution | up to 2 years of age
  pulmonary hypertension will be collected from medical chart review.

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Fetal Care Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No